CLINICAL TRIAL: NCT06476197
Title: A Single Center, Single Arm, Prospective , Exploratory Clinical Trial to Evaluate the Validity, Safety and Efficacy of SAT-003 in Cancer Cachexia Patients Discontinued Chemotherapy Who Had Diagnosed With Solid Cancer
Brief Title: Exploratory Trial of SAT-003 in Cancer Cachexia Patients With Discontinued Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S-Alpha Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAT003-KP-001
Record Dates: First submitted 2024-05-27; First posted 2024-06-26 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Cancer Cachexia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SAT-003 Treatment arm(Single arm) (Experimental): Arm Name: SAT-003 Treatment Arm
  Intervention:
  * Type: Software Device (Rehabilitation Medicine Software, E10000, Class 2 Medical Device)
  * Name: SAT-003
  * Details: Participants will use the SAT-003 software daily 10 mins at most/ for 12 weeks. Specific usage instructions and session duration will be provided according to the protocol.
  Arm Description: This is a single-arm, prospective exploratory clinical trial. All participants, who are patients with cancer cachexia diagnosed with solid tumors and having discontinued chemotherapy, due to cancer cachexia, will receive the investigational medical device, SAT-003. The primary objective of this arm is to evaluate the feasibility of safety, and preliminary efficacy of SAT-003. Participants will undergo specified assessments at Baseline, Week 6, Week 12, and Week 24 to monitor their progress and potential adverse events. No control group or comparative intervention will be administered in this study.
  Interventions: Device: SAT-003

INTERVENTIONS:
Device: SAT-003 — Device: SAT-003(Software) Using SAT-003 for 12 weeks

SUMMARY:
This clinical trial aims to evaluate the feasibility of 'SAT-003' as well as its exploratory safety and efficacy in patients with cancer cachexia who have been diagnosed with solid tumors and have discontinued anticancer treatment.

DETAILED DESCRIPTION:
Cancer cachexia, characterized by weight loss, anorexia, and muscle wasting, is a metabolic imbalance resulting from impaired endocrine function. Unlike simple hunger or loss of appetite, cancer cachexia leads to a reduction in weight and skeletal muscle metabolism despite normal food intake, progressively weakening the body's overall function. Many cancer patients experience this condition, which can increase resistance to cancer treatment, worsen overall health, and diminish quality of life, often leading to the discontinuation of therapy. Cancer cachexia is a common complication in cancer patients and is associated with high mortality rates. Despite ongoing research, no effective treatment for cancer cachexia has been identified, and current therapies targeting appetite improvement or nutritional support often fail to effectively address the full spectrum of symptoms. SAT-003 has been developed to alleviate the symptoms of cancer cachexia and facilitate the resumption of cancer treatment. This single-center, single-arm, prospective feasibility clinical trial aims to evaluate the feasibility, safety, and effectiveness of SAT-003 in patients with cancer cachexia who have been diagnosed with solid tumors and discontinued chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 19 years and older
2. Cancer cachexia patients diagnosed with solid tumors and whose anticancer treatments (surgery, radiation therapy, anticancer drugs, or chemotherapy) have been discontinued. (Diagnosis criteria for cancer cachexia include: experiencing a weight loss of 5% or more over the past 6 months, having a BMI below 20 with a weight loss exceeding 2%, or having a skeletal muscle index indicative of sarcopenia (for males < 7.26 kg/m^2; for females < 5.45 kg/m^2) with a weight loss exceeding 2%
3. between 20 and 70 points of KPS score
4. Capable of holding and raising a smartphone with the treatment application installed
5. Capable of either listening or viewing, and able to move parts of their body
6. Capable of using a smartphone and application by themselves or with assistance from caregiver or guardian (In the latter case, the availability of assistance from a caregiver or guardian shoud be confirmed.)

Exclusion Criteria:

1. have pledged discontinue further anticancer treatment
2. Those whose chemotherapy or radiation therapy has already been confirmed prior to enroll
3. lack the cognitive ability to understand and adhere the instructions

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-11 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Change in Karnofsky Performance Status(KPS)score | Baseline, 6weeks, 12weeks, 18weeks, 24weeks
  The change in the Karnofsky Performance Status (KPS) score was evaluated from Baseline (Visit 2) to Week 6 (Visit 5) and Week 12 (Visit 8) post-treatment, and also from Week 6 (Visit 5) to Week 12 (Visit 8) post-treatment.
  The KPS score is a scale used to assess a patient's recovery process to daily living after treatment. A score of 0 indicates the worst, non-functional state, while 100 represents a normal state.
Change in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) score | Baseline, 6weeks, 12weeks, 18weeks, 24weeks
  The change in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) score was evaluated from Baseline (Visit 2) to Week 6 (Visit 5) and Week 12 (Visit 8) post-treatment, and also from Week 6 (Visit 5) to Week 12 (Visit 8) post-treatment.
  The EORTC QLQ-C30 is a 30-item questionnaire composed of three domains: global health status/quality of life, functional scales, and symptom scales. The global health status is assessed by 2 items, while the functional scales consist of 15 items evaluating physical, role, cognitive, emotional, and social functioning. The symptom scales include 2-3 items for fatigue, pain, and nausea/vomiting, and single items for dyspnea, appetite loss, sleep disturbance, constipation, diarrhea, and financial difficulties. Scores range from 0 to 100. Higher scores for global health status and functional scales, and lower scores for symptom scales, indicate a better quality of life.
Chagne in Korean Modified Barthel Index (KBMI) Score | Baseline, 6weeks, 12weeks, 18weeks, 24weeks
  The change in the Korean Modified Barthel Index (KMBI) score was evaluated from Baseline (Visit 2) to Week 6 (Visit 5) and Week 12 (Visit 8) post-treatment, and also from Week 6 (Visit 5) to Week 12 (Visit 8) post-treatment.
  The K-MBI is an indicator used to assess a patient's performance in activities of daily living (ADL). A score of 100 represents a normal state requiring no assistance with daily activities, and the score decreases as more assistance is needed (refer to Appendix 4. Korean version of Modified Barthel Index Questionnaire).
Change in Grip Strength(Hand grip, Pinch grip, Lateral prehension, Three jaw chuck) (lbs) | Baseline, 6weeks, 12weeks, 18weeks, 24weeks
  The change in Grip Strength (Hand grip, Pinch grip, Lateral prehension, Three jaw chuck) were evaluated from Baseline (Visit 2) to Week 6 (Visit 5) and Week 12 (Visit 8) post-treatment, and also from Week 6 (Visit 5) to Week 12 (Visit 8) post-treatment. *Handgrip strength was measured using a JAMAR Hydraulic Hand Dynamometer, and pinch strength was measured using a JAMAR Hydraulic Pinch Gauge.
  Hand grip, Pinch grip, Lateral prehension, and Three jaw chuck are measured using a handgrip dynamometer and pinch gauge. Before performing each item, the assessor explains and demonstrates the task to the subject. The subject attempts each hand three times, with a rest period after each attempt. The results are evaluated as the average value for each hand.
Rate of Change (%) in Grip Strength(Hand grip, Pinch grip, Lateral prehension, Three jaw chuck) (lbs) | Baseline, 6weeks, 12weeks, 18weeks, 24weeks
  The change rate in Grip Strength (Hand grip, Pinch grip, Lateral prehension, Three jaw chuck) were evaluated from Baseline (Visit 2) to Week 6 (Visit 5) and Week 12 (Visit 8) post-treatment, and also from Week 6 (Visit 5) to Week 12 (Visit 8) post-treatment. *Handgrip strength was measured using a JAMAR Hydraulic Hand Dynamometer, and pinch strength was measured using a JAMAR Hydraulic Pinch Gauge.
  Hand grip, Pinch grip, Lateral prehension, and Three jaw chuck are measured using a handgrip dynamometer and pinch gauge. Before performing each item, the assessor explains and demonstrates the task to the subject. The subject attempts each hand three times, with a rest period after each attempt. The results are evaluated as the average value for each hand.
Change in Lean Body Mass(LBM) and Rate of LBM Change (%) | Baseline, 6weeks, 12weeks, 18weeks, 24weeks
  The change and change rate in Lean Body Mass (LBM) were evaluated from Baseline (Visit 2) to Week 6 (Visit 5) and Week 12 (Visit 8) post-treatment, and also from Week 6 (Visit 5) to Week 12 (Visit 8) post-treatment. *LBM is measured according to the institution's standard procedures using Dual Energy X-ray Absorptiometry (DEXA).
Survival Rate (%) at 24 weeks | Baseline, 24weeks
  The proportion of surviving subjects who survived up to 24 weeks after enrollment is evaluated.
  To assess the proportion of subjects surviving to 24 weeks after the date of enrollment.
Chemotherapy Resumption Rate(%) | 12 weeks, 24weeks
  The proportion of patients who resumed chemotherapy and the time (days) elapsed until chemotherapy resumption are evaluated at Week 12 (Visit 8) and Week 24 (Visit 9) post-treatment
Chemotherapy Resumption period(days) | 24weeks
  The evaluate the duration from application SAT-003 to resumption of chemotherapy.

SECONDARY OUTCOMES:
Adherence Assessment During the Treatment Period | Baseline, Week12, through study completion, an average of 24 weeks
  Adherence to device use, measured by the number of sessions performed within the specified period, is evaluated weekly from Baseline (Visit 2) to Week 12 (Visit 8) post-treatment.
Change in Number of External Activity Performances | Baseline, Week12, through study completion, an average of 24 weeks
  The change in external activity performance, measured weekly using the investigational medical device, is evaluated from Baseline (Visit 2) to Week 12 (Visit 8) post-treatment. The change in external activity is calculated by comparing the initial number of activity performances within a session to the last data point of the session week.

OTHER OUTCOMES:
Adverse Events | through study completion, an average of 24 weeks
  Adverse events are classified into those occurring before the application of the investigational medical device and those occurring after its application (referred to as Treatment Emergent Adverse Events, TEAEs). Adverse events that occurred before the application of the investigational medical device is recorded as pre-treatment adverse events but is excluded from the adverse event analysis. In other words, the adverse event analysis focused solely on TEAEs. However, signs and symptoms arising from the progression of the underlying disease (cancer and cancer cachexia) is not considered adverse events or serious adverse events. Furthermore, for fluctuations in symptoms commonly occurring due to the underlying disease, the investigator determine whether they constituted an adverse event after considering the patient's health status and other factors.

CONTACTS AND LOCATIONS:
Overall Officials: Dalyong Kim, M.D., Ph.D, Principal Investigator — DongGuk University
Locations (1):
- Dongguk University Ilsan Hospital, Ilsan, Gyeonggi-do, South Korea